CLINICAL TRIAL: NCT05332665
Title: Anterior Segment Optical Coherence Tomography Evaluation of Iridocorneal Angle of Patients of Angle Closure Glaucoma After Phacoemulsification and YAG Laser Iridotomy, Comparative Study
Brief Title: AS-OCT Evaluation of Iridocorneal Angle of Patients of Angle Closure Glaucoma After Phacoemulsification
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mohamed Salah, Principal Investigator, Minia University
Other Study IDs: AS-OCT in ACG
Record Dates: First submitted 2022-03-28; First posted 2022-04-18 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Glaucoma, Angle-Closure
MeSH Terms: conditions — Glaucoma, Angle-Closure

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Angle opening distance (AOD): The AOD measured as perpendicular distance between anterior iris surface and point at trabecular meshwork at 500 μm anterior to the scleral spur
  Interventions: Device: AS-OCT; Procedure: YAG laser PI
- Trabecular iris space area (TISA) 500: TISA 500 was measured as an area bounded anteriorly by the AOD 500, posteriorly by a line drawn from the scleral spur perpendicular to the plane of the inner scleral wall to the opposing iris, superiorly by the inner corneoscleral wall, and inferiorly by the iris surface
  Interventions: Device: AS-OCT; Procedure: YAG laser PI
- Anterior chamber depth (ACD): The ACD was measured as the perpendicular distance from the corneal endothelium at the corneal apex to the anterior lens surface
  Interventions: Device: AS-OCT; Procedure: YAG laser PI

INTERVENTIONS:
Device: AS-OCT — Anterior segment optical coherence tomography (AS OCT) is an imaging device that can acquire an anterior segment image using a noncontact method with the patient in a sitting position. This device provides reproducible and quantitative measurements of the AC angle and other anterior segment parameters.
Procedure: YAG laser PI — medical procedure which uses a laser device to create a hole in the iris, thereby allowing aqueous humor to traverse directly from the posterior to the anterior chamber and, consequently, relieve a pupillary block

SUMMARY:
Evaluation of the effect of phacoemulsification and YAG Laser peripheral iridotomy on the anterior chamber angle anatomic parameters in PACG eyes, using anterior segment optical coherence tomography (SS ASOCT) device

DETAILED DESCRIPTION:
The recent treatment of ACG is phacoemulsification in patients of acute attack with YAG laser iridotomy in the other eye.

The AS-OCT will be used for evaluation of the angle of the anterior chamber parameters in both eyes after phacoemulsification and YAG laser peripheral iridotomy.

Follow up of AS-OCT will be done 1,3,6 months after surgery and we will compare results in each eye and between both eyes.

.

ELIGIBILITY:
Inclusion Criteria:

* patients with acute attack of angle closure glaucoma in one eye.
* Patients fit for phacoemulsification

Exclusion Criteria:

* 1- Patients with history of any intraocular surgery. 2- Patients with history of refractive surgery. 3- Patients with diabetic retinal vasculopathy or retinal detachment. 4- Patients with chronic angle closure glaucoma, open angle glaucoma or 2ry glaucoma

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with acute attack of ACG with phacoemulsification in this eye with YAG laser PI in the other eye
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2022-01-11 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
IOP | up to 6 months
  mmhg

SECONDARY OUTCOMES:
Corneal endothelial count | up to 6 months
  CD per mm2

CONTACTS AND LOCATIONS:
Overall Officials: mohamed Salah, Principal Investigator — Minia faculty of medicine
Locations (1):
- mohamed Mahmoud, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Not decided